CLINICAL TRIAL: NCT03823794
Title: The Epidemiology of Atopic Dermatitis, Associated Comorbidities, and Treatment Patterns in the United Kingdom (UK)
Brief Title: Trends in the Epidemiology and Treatment of Atopic Dermatitis in the United Kingdom (UK)
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry); Oxford Royal College of General Practitioners Research and Surveillance Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: P002
Record Dates: First submitted 2019-01-17; First posted 2019-01-30 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis Eczema; Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active atopic dermatitis: People fulfilling the diagnostic criteria for active atopic dermatitis during the calendar year 2018, and meeting the inclusion criteria and registered with one of the study practices for one or more years during the study period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational analysis of usual care only

SUMMARY:
Atopic dermatitis (AD), commonly called eczema, is one of the most frequently occurring skin conditions. It is estimated to affect around one fifth of children in developed countries and is also becoming increasingly common in less developed countries. Exact estimates of how common eczema is, vary considerably and there has not been an in-depth analysis of the number of people with eczema in the UK. It is also unclear which groups of people are most affected and which treatment options are being used.

Most people with eczema are managed by their general practitioner (GP) with only a few people requiring specialist care. GP records therefore provide an excellent opportunity to explore how common eczema is and which treatments are being used currently.

DETAILED DESCRIPTION:
Objective

The study aims to describe the health care resource utilisation of patients with active AD in terms of prescription use, primary care appointments, and specialist referrals.

Method This study will define AD cases using a previously validated algorithm for case identification use clinical codes form primary care in the UK (Read codes). The study will analyse a cohort of prevalent active AD cases over a one year period (2018). The annual use of topical and oral medications used for the treatment of AD, primary care appointments, and specialist referrals will be reported.

ELIGIBILITY:
Inclusion Criteria:

* All paediatric and adult patients registered with an Royal College of General Practitioners (RCGP) Research and Surveillance Centre (RSC) contributing GP practice during the study period (2008-2018) and with at least one year of follow-up.

Exclusion Criteria:

* The presence of psoriasis, photodermatitis, or ichthyosis

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with atopic dermatitis identified from routinely collected healthcare records using a validated algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 148166 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data Ltd
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data (IPD) can be made available to bone fide researchers subject to appropriate checks and approvals made by Momentum Data, the RCGP RSC, and the University of Surrey and subject to the completion of information governance training.
Supporting Information: Study Protocol
Time Frame: There is no pre-specified time-frame for data availability; this will be considered on an individual basis for each request.
Access Criteria: As above

REFERENCES:
- [Derived] de Lusignan S, Alexander H, Broderick C, Dennis J, McGovern A, Feeney C, Flohr C. The epidemiology of eczema in children and adults in England: A population-based study using primary care data. Clin Exp Allergy. 2021 Mar;51(3):471-482. doi: 10.1111/cea.13784. Epub 2020 Nov 26. PMID 33179341
- [Derived] de Lusignan S, Alexander H, Broderick C, Dennis J, McGovern A, Feeney C, Flohr C. Patterns and trends in eczema management in UK primary care (2009-2018): A population-based cohort study. Clin Exp Allergy. 2021 Mar;51(3):483-494. doi: 10.1111/cea.13783. Epub 2020 Nov 23. PMID 33176023
- [Derived] de Lusignan S, Alexander H, Broderick C, Dennis J, McGovern A, Feeney C, Flohr C. Epidemiology and management of atopic dermatitis in England: an observational cohort study protocol. BMJ Open. 2020 Sep 16;10(9):e037518. doi: 10.1136/bmjopen-2020-037518. PMID 32938595

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Atopic Dermatitis: People fulfilling the diagnostic criteria for active atopic dermatitis (AD) during the calendar year 2018. Primary outcomes conducted within this single arm.
  No intervention: Observational analysis of usual care only
Period: Overall Study
Arm/Group | Active Atopic Dermatitis
Started | 148166
Completed | 148166
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Atopic Dermatitis: People fulfilling the diagnostic criteria for active atopic dermatitis during the calendar year 2018. Primary outcomes conducted within this single arm.
  No intervention: Observational analysis of usual care only
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Age, Customized [Count of Participants; unit: Participants]
  Age Group: <2 | 7230
  Age Group: 2-11 | 34074
  Age Group: 12-17 | 12476
  Age Group: 18-49 | 37995
  Age Group: >=50 | 56391
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81357
  Male | 66809
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 87717
  Ethnicity: Asian | 14980
  Ethnicity: Black | 5799
  Ethnicity: Mixed | 2808
  Ethnicity: Other | 1234
  Ethnicity: Missing | 35628
IMD quintile [Count of Participants; unit: Participants] — Index of Multiple Deprivation (IMD) is a UK national deprivation measure of deprivation which is based on the patient postcode. IMD has been stratified into quintiles with IMD 1 representing most deprived and IMD 5 being the least deprived.
  Participants
    1 (most deprived) | 26454
    2 | 25520
    3 | 26445
    4 | 31426
    5 (least deprived) | 36467
    Missing | 1854
Rural-urban classification [Count of Participants; unit: Participants]
  Urban | 117466
  Rural | 29005
  Missing | 1695

OUTCOME MEASURES:

1. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Emollients and Soap Substitutes
Description: Proportion of the arm/group receiving at least one prescription for emollients and soap substitutes.
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 76095

2. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Mild Topical Corticosteroids (TCS)
Description: Proportion of the arm/group receiving at least one prescription for mild topical corticosteroids (atopic dermatitis related treatment)
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 40478

3. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Moderate Topical Corticosteroids (TCS)
Description: Proportion of the arm/group receiving at least one prescription for moderate topical corticosteroids (an atopic dermatitis related treatment)
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 19575

4. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Potent Topical Corticosteroids (TCS)
Description: Proportion of the arm/group receiving at least one prescription for potent topical corticosteroids (an atopic dermatitis related treatment)
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 34997

5. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Very Potent Topical Corticosteroids (TCS)
Description: Proportion of the arm/group receiving at least one prescription for very potent topical corticosteroid (an atopic dermatitis related treatment)
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 6478

6. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Topical Calcineurin Inhibitors (TCI)
Description: Proportion of the arm/group receiving at least one prescription for a topical Calcineurin Inhibitor (an atopic dermatitis related treatment)
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 2683

7. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Topical Antimicrobials
Description: Proportion of the arm/group receiving at least one prescription for topical antimicrobials.
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 19378

8. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Antihistamin
Description: Proportion of the arm/group receiving at least one prescription for antihistamin.
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 29041

9. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Systemic Immuno-modulatory Therapy
Description: Proportion of the arm/group receiving at least one prescription for Systemic immuno-modulatory therapy
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 2785

10. Primary Outcome: Prescription Rates for Atopic Dermatitis Related Treatments: Oral Corticosteroids
Description: Proportion of the arm/group receiving at least one prescription for oral corticosteroids
Time Frame: Jan - Dec 2018 inclusive
Measure: Count of Participants; unit: Participants
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Participants | 12087

11. Primary Outcome: Specialist Referrals
Description: Specialist dermatology referral rate in 2018
Time Frame: Jan - Dec 2018 inclusive
Measure: Number (95% Confidence Interval); unit: Referrals per 100 person-years
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Referrals per 100 person-years | 5.0 [4.9 to 5.1]

12. Primary Outcome: Primary Care Referrals
Description: Annual rate of primary care consultations in 2018
Time Frame: Jan - Dec 2018 inclusive
Measure: Number (95% Confidence Interval); unit: Consultations per 100 person-years
Arm/Group | Active Atopic Dermatitis
Number analyzed (Participants) | 148166
Consultations per 100 person-years | 112.0 [111.5 to 112.6]

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for the study.
Arm/Group | Active Atopic Dermatitis
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT03823794/Prot_SAP_001.pdf